CLINICAL TRIAL: NCT02481752
Title: The Effect of AAT Training in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2015-02-0023
Record Dates: First submitted 2015-06-17; First posted 2015-06-25 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Tobacco Use
Keywords: Tobacco Use; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AAT Training Group (Experimental): Individuals in this condition will receive four sessions of AAT training in which they are instructed to approach (pull the joystick) images tilted to the right and avoid (push the joystick) images tilted to the left. They will be told that the training may weaken automatic cigarette-approach and strengthen automatic cigarette-avoidance. Furthermore, they will be told that the opposite effect will be true for the stimuli not related to cigarettes (i.e., the positive stimuli).
  Interventions: Other: Approach Avoidance Training
- SHAM Training Group (Sham Comparator): Individuals in this condition will receive four sessions of SHAM training in which they are instructed to approach (pull the joystick) images tilted to the right and avoid (push the joystick) images tilted to the left. They will be told that the purpose of the training is to improve control over these automatic tendencies and that following the training sessions, they will easily be able to push or pull the stimuli regardless of content.
  Interventions: Other: SHAM Training

INTERVENTIONS:
Other: Approach Avoidance Training — The Approach Avoidance Task (AAT) used for this experiment is an implicit, computerized paradigm in which participants respond to visually presented pictures on a computer screen displaying either 1) smoking-related images or 2) positive images, by pulling a joystick either towards their body (approach movement) or pushing it away from their body (avoidance movement). By pulling the joystick towards their body, the picture grows in size; by pushing the joystick away, the picture shrinks and then disappears from the screen. Participants are instructed to pull upon seeing an image tilted to the right and to push upon seeing a left-tilt image, while ignoring the image content and responding as quickly and as accurately as possible.
  Arms: AAT Training Group
Other: SHAM Training
  Arms: SHAM Training Group

SUMMARY:
The purpose of this research study is to investigate the effect of a brief computer task (Approach Avoidance Task) on smoking cessation. The investigators will use a novel training protocol that works to target automatic thoughts and tendencies that occur outside of conscious control. Previous research suggests that these automatic tendencies may have a direct effect on certain health behaviors- like continuing to smoke despite having previous quit attempts.

The investigators hypothesize that individuals in the AAT training condition will evidence a greater decrease in reaction times to avoid smoking-related stimuli & approach positive stimuli relative to those in the control condition. The investigators also expect that individuals in the AAT condition will exhibit superior outcomes on several quit-related variables as evidenced by an increase in motivation to quit smoking, an increase in number of days abstinent following a self-guided quit attempt, an increase in self-efficacy, and a decrease in urge to smoke compared to those in the SHAM training condition.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18-65 capable of providing informed consent
* Willing and able to provide informed consent, attend all study visits, and comply with the protocol
* Daily smoker for at least 6 months
* Currently smoke an average of at least 8 cigarettes per day
* Report a motivation to quit smoking of at least 5 on a 10-point scale
* Interest in making a serious quit attempt within the next month (without professional assistance or nicotine therapy)
* Have not decreased their number of cigarettes by more than half in the last six months

Exclusion Criteria:

* Visual or hand-motoric impairments
* Current use of nicotine replacement therapy
* Current use of tobacco products other than cigarettes
* Insufficient command of the English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reaction Time on Approach Avoidance Task | 2 weeks
  The time between the start of the trial and the picture disappearing from the screen will be recorded. The investigators will look at the change in response times for each individual. The investigators hypothesize that there will be a greater decrease in reaction time for those in the AAT training group.

SECONDARY OUTCOMES:
Motivation to Quit Smoking as assessed by having participants rate their motivation to quit smoking on a scale of 1 to 10 (1 being not motivated at all and 10 being extremely motivated to quit). | 2 weeks
  The investigators expect that individuals in the AAT training condition will have a greater motivation to quit smoking relative to those in the SHAM condition.
Number of Days Abstinent as assessed by daily cigarette count during a self-guided quit attempt. | 2 weeks
  The investigators hypothesize that individuals in the AAT training condition will be more likely to have a greater number of days abstinent following Quit Day relative to those in the SHAM condition.
Self Efficacy as assessed by the Relapse Situation Self-Efficacy questionnaire. | 2 weeks
  The investigators expect to see a greater increase in self-efficacy for the AAT training group relative to the SHAM training group.
Urge to Smoke as assessed by the QSU-brief (Questionnaire of Smoking Urges). | 2 weeks
  The investigators hypothesize that individuals in the AAT training condition will evidence a greater decrease in urge to smoke relative to those in the SHAM condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jasper A Smits, Ph.D., Principal Investigator — University of Texas at Austin; Scarlett O Baird, B.A., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States